CLINICAL TRIAL: NCT04438772
Title: Effect of LPEC Compared With a Sham Procedure in the General Anesthesia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Benjamin Javillier, Principal Investigator, University of Liege
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: LPEConditions
Record Dates: First submitted 2020-06-15; First posted 2020-06-19 (Actual); Last update posted 2020-06-19 (Actual); Status verified 2020-06

CONDITIONS: Intubation;Difficult

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LPEC (Experimental)
  Interventions: Other: Check the condition of intubation with LPEC compared with a sham procedure in the general anesthesia
- Sham procedure (Sham Comparator)
  Interventions: Other: Check the condition of intubation with LPEC compared with a sham procedure in the general anesthesia

INTERVENTIONS:
Other: Check the condition of intubation with LPEC compared with a sham procedure in the general anesthesia — Intubation with Left Paratracheal Esophagus Compression (LPEC) or sham procedure and evaluation of intubation's condition

SUMMARY:
Check the condition of intubation with LPEC compared with a sham procedure in the general anesthesia

ELIGIBILITY:
Inclusion Criteria:

* Intubation

Exclusion Criteria:

* ENT neoplasia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2020-10-01 (Estimated); Study Completion 2020-11-01 (Estimated)

PRIMARY OUTCOMES:
Cormack score | During laryngoscopy
  from 0 to 4

SECONDARY OUTCOMES:
Time to intubation | During laryngoscopy

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Javillier, MD, Principal Investigator — University of Liege
Locations (1):
- Javillier, Liège, Belgium